CLINICAL TRIAL: NCT01201642
Title: Prednisone Acetate and Acupuncture for the Treatment of Facial Neuritis: a Multiple Center, Comparative Effectiveness Research in China
Brief Title: Prednisone and Acupuncture for the Treatment of Facial Neuritis: a Multiple Center, CER in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XijingNeuro-2010
Record Dates: First submitted 2010-08-30; First posted 2010-09-14 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Bell's Palsy
Keywords: Bell's palsy; Prednisolone; acupuncture
MeSH Terms: conditions — Bell Palsy | interventions — Prednisolone; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Prednisolone (Experimental): Prednisolone as 5 mg tablets will be given within 72 h after onset of Bell's palsy as a single dose of 40 mg daily for 5 days; the dose will then be reduced by 10 mg per 5 day, with a total treatment time of 20 days.
  Interventions: Drug: Prednisolone
- Acute stage acupuncture (Experimental): Accept acupuncture therapy within 10days after onset of Bell's palsy, do not accept prednisolone therapy. The acupuncture points used were Dicang (ST4), Jiache (ST6), Yangbai (GB14), Xiaguan (ST7), Taiyang (EX-HN5), Quanliao (SI18) and Yifeng (TE17) on the affected side, and Hegu (LI4) bilaterally. For acute stages acupuncture, shallow puncturing is used at facial acupoints and routine puncturing is used at other acupoints within 72 h after onset of Bell's palsy. Yifeng (TE17), Hegu (LI4) are punctured 0.5-1.0 cun, the others are punctured 0.1-0.3 cun. and the needles were retained for 30 minutes, once a day, five times a week, for a total period of four weeks.
  Interventions: Device: acupuncture
- Prednisolone + acute stage acupuncture (Experimental): Accept prednisolone and acupuncture therapy within 10days after onset of Bwll's palsy. Prednisolone used as same as the Arm of Prednisolone. The acupuncture points used as same as the Arm of Acute stage acupuncture.
  Interventions: Drug: Prednisolone; Device: acupuncture
- Resting stage acupuncture (Experimental): Accepted acupuncture therapy after 10 days of the onset of Bell's palsy. The acupuncture points used were Dicang (ST4), Jiache (ST6), Yangbai (GB14), Xiaguan (ST7), Taiyang (EX-HN5), Quanliao (SI18) and Yifeng (TE17) on the affected side, and Hegu (LI4) bilaterally. Penetrative needling is used from Dicang (ST4) to Jiache (ST6) and from Taiyang (EX-HN5) to Quanliao (SI18) 2-3 cun, and routine puncturing is used at other acupoints 7 d after enrolment. Filiform needles (33 - 49.5 mm, 0.32 mm) will be used with moderate stimulation to get an acupuncture sensation, and the needles were retained for 30 minutes, once a day, five times a week, for a total period of four weeks.
  Interventions: Device: acupuncture
- Prednisolone + resting stage acupuncture (Experimental): Accept prednisolone and acupuncture therapy more than 10days after onset of Bwll's palsy. Prednisolone used as same as the Arm of Prednisolone. The acupuncture points used as same as the Arm of Resting stage acupuncture.
  Interventions: Drug: Prednisolone; Device: acupuncture
- Other treatment (Other): Do not accept neither prednisolone nor acupuncture therapy. The therapy accepted is different from the five Arms Previously.
  Interventions: Other: other treatment

INTERVENTIONS:
Drug: Prednisolone — Prednisolone as 5 mg tablets will be given as a single dose of 40 mg daily for 10 days; the dose will then be reduced by 10 mg per 5 day, with a total treatment time of 20 days.
  Arms: Prednisolone; Prednisolone + acute stage acupuncture; Prednisolone + resting stage acupuncture
Device: acupuncture — The acupuncture points used were Dicang (ST4), Jiache (ST6), Yangbai (GB14), Xiaguan (ST7), Taiyang (EX-HN5), Quanliao (SI18) and Yifeng (TE17) on the affected side, and Hegu (LI4) bilaterally. For acute stages acupuncture, shallow puncturing is used at facial acupoints and routine puncturing is used at other acupoints. For resting stage acupuncture, penetrative needling is used from Dicang (ST4) to Jiache (ST6) and from Taiyang (EX-HN5) to Quanliao (SI18) 2-3 cun, and routine puncturing is used at other acupoints. Filiform needles (33 - 49.5 mm, 0.32 mm) will be used with moderate stimulation to get an acupuncture sensation, and the needles were retained for 30 minutes, once a day, five times a week, for a total period of four weeks.
  Arms: Acute stage acupuncture; Prednisolone + acute stage acupuncture; Prednisolone + resting stage acupuncture; Resting stage acupuncture
Other: other treatment — common medicine or other physical treatment which are different from those 5 Arms Previously.
  Arms: Other treatment

SUMMARY:
The aim of this study is to compare the effects of prednisolone and staging acupuncture in the recovery of the affected facial nerve, and to verify that whether in combination with staging acupuncture is more effective than prednisolone alone for Bell's palsy in a large number of patients.

DETAILED DESCRIPTION:
Patients will be recruited between Sep, 2010, and Dec, 2014. Baseline assessments before the start of treatment include neurological examination, grading of facial function, measurement of ipsilateral pain, documentation of concurrent medication.

These patients are assigned to receive one of the following treatment groups, i.e. 1)the hormone group: oral hormone drugs, do not accept acupuncture treatment; 2)acupuncture group: using acupuncture therapy, do not accept oral hormone therapy; 3)hormone-acupuncture combined treatment group: receive oral hormone and acupuncture therapy at the same time; 4)other treatment group: other treatment in addition to the above 3 groups of treatment abroad. The secondary factor grouping (subgroup): According to the different time of treatment after the onset of disease, the acupuncture group and the hormone- acupuncture combined treatment group can be divided into Type Ⅰ subgroup (patients receive acupuncture within 10 days of the onset of disease) and Type II subgroups (patients receive acupuncture after 10 days of the onset of disease). The primary outcome is the time to complete recovery of facial function, assessed by Sunnybrook system and House-Brackmann scale. The secondary outcomes include the incidence of ipsilateral pain in the early stage of palsy (and the duration of this pain), the proportion of patients with severe pain, the occurrence of synkinesis, facial spasm or contracture, and the severity of residual facial symptoms during the study period.

ELIGIBILITY:
Inclusion Criteria:

* involvement of unilateralfacial nerve paralysis only
* aged between 18 and 75 years old
* period of onset of facial paralysis within 72h

Exclusion Criteria:

* pregnancy
* breastfeeding
* being a woman of child bearing age who is unwilling to use contraceptives during the medication period
* other neurological diseases
* diabetes
* badly controlled hypertension
* current or a history of serious heart disease
* history of renal or hepatic disease
* gastric or duodenal ulcer
* history of glaucoma
* acute otitis or history of ipsilateral chronic otitis
* history of tuberculosis, history of immunodeficiency syndromes
* recent head injury, psychiatric disease, or any other condition that is at risk of being inﬂuenced by the study medication or that might have affected completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-12 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of Facial function | 10days, 1 month, 2 months, 3months, 4months, 6months
  Facial function will be assessed at all visits with two grading systems（ The Sunnybrook system and The House-Brackmann scale ）.If recovery is complete (Sunnybrook scale score of 100 points), the next follow-up will be at 6 months.

SECONDARY OUTCOMES:
Neurology examination | 10days, 1 month, 2 months, 3months, 4months, 6months
  Pain around the ear, in the face, or in the neck will be registered on a visual analogue scale that ranges from 0 to 10 points, where 0 is no pain and 10 very severe pain. Occurrence of facial spasm or contracture and synkinesia in the different treatment arms at any time will be observed and recorded.
registration of ipsilateral pain | 10days, 1 month, 2 months, 3months, 4months, 6months
  Pain around the ear, in the face, or in the neck will be registered on a visual analogue scale that rangs from 0 to 10 points, where 0 is no pain and 10 very severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, MD, Study Director — the Department of Neurology , Xijing Hospital; Feng Xia, MD, Study Chair — the Department of Neurology , Xijing Hospital
Locations (1):
- the Department of Neurology , Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Xia F, Han J, Liu X, Wang J, Jiang Z, Wang K, Wu S, Zhao G. Prednisolone and acupuncture in Bell's palsy: study protocol for a randomized, controlled trial. Trials. 2011 Jun 21;12:158. doi: 10.1186/1745-6215-12-158. PMID 21693007